CLINICAL TRIAL: NCT07344467
Title: Effect of Oral Melatonin Versus Oral Pregabalin on Postoperative Pain and Anxiety Following Spine Surgery: A Prospective, Randomized Controlled Trial
Brief Title: Oral Melatonin Versus Oral Pregabalin on Postoperative Pain and Anxiety Following Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Hamdy Said Ayad, Assistant lecturer of Anesthesia, Surgical Intensive Care and Pain Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36265MD429/6/25
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Oral; Melatonin; Pregabalin; Postoperative Pain; Anxiety; Spine Surgery
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders | interventions — Melatonin; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Control Group) (Placebo Comparator): Patients will be receive one oral placebo capsule the evening before surgery, one oral placebo capsule 2 hours prior to surgery, and one oral placebo capsule in the morning and one in the evening for 3 consecutive days postoperatively.
  Interventions: Other: Placebo capsule
- Group M (Melatonin Group) (Experimental): Participants will receive one 5 mg oral melatonin capsule the evening before surgery, one 5 mg oral melatonin capsule 2 hours prior to surgery, and one oral placebo capsule in the morning, and one 5 mg oral melatonin capsule in the evening, daily for 3 consecutive days postoperatively.
  Interventions: Drug: Melatonin capsule
- Group P (Pregabalin Group) (Experimental): Participants will receive one 75 mg oral pregabalin capsule the evening before surgery, one 75 mg oral pregabalin capsule 2 hours prior to surgery, and one 75 mg oral pregabalin capsule in the morning, and another in the evening, daily for 3 consecutive days postoperatively.
  Interventions: Drug: Pregabalin capsule

INTERVENTIONS:
Other: Placebo capsule — Patients will be receive one oral placebo capsule the evening before surgery, one oral placebo capsule 2 hours prior to surgery, and one oral placebo capsule in the morning and one in the evening for 3 consecutive days postoperatively.
  Arms: Group C (Control Group)
Drug: Melatonin capsule — Participants will receive one 5 mg oral melatonin capsule the evening before surgery, one 5 mg oral melatonin capsule 2 hours prior to surgery, and one oral placebo capsule in the morning, and one 5 mg oral melatonin capsule in the evening, daily for 3 consecutive days postoperatively.
  Arms: Group M (Melatonin Group)
Drug: Pregabalin capsule — Participants will receive one 75 mg oral pregabalin capsule the evening before surgery, one 75 mg oral pregabalin capsule 2 hours prior to surgery, and one 75 mg oral pregabalin capsule in the morning, and another in the evening, daily for 3 consecutive days postoperatively.
  Arms: Group P (Pregabalin Group)

SUMMARY:
This study aims to compare the efficacy of using Melatonin versus Pregabalin on postoperative pain and anxiety after spine surgeries.

DETAILED DESCRIPTION:
Spine surgery is one of the most common procedures performed every day which is associated with intense pain in the postoperative period, mostly in the first few days after surgery. Effective pain management leads to improved functional outcomes, early ambulation, prevention of chronic pain and early discharge.

Melatonin is neurohormone mainly secreted from the pineal gland by the suprachiasmatic nucleus. This neurohormone possesses a circadian secretion pattern and regulates the biological clock; it also offers antiemetic, analgesic, and anxiolytic effects.

Pregabalin is a structural analogue of gamma-aminobutyric acid that acts as a potent ligand for alpha 2-delta subunits of the voltage-gated calcium channels in the nervous system. Such action results in a reduction in the depolarization-induced influx of calcium, hence a reduction in the release of excitatory neurotransmitters including glutamate, noradrenaline, dopamine, and serotonin.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21-60 years old.
* Both sexes.
* Patients of American Society of Anesthesiologists (ASA) physical status I & II.
* Undergoing elective spine surgery.

Exclusion Criteria:

* Patient refusal.
* History of allergic reactions to melatonin or pregabalin.
* Patients with cardiovascular disease (ischemic heart disease, Heart Failure, Arrythmia, Heart Block).
* Patients with kidney disease with (plasma creatinine level > 1.5mg/dl).
* Patients with liver disease with (aspartate transaminase, alanine transaminase, and bilirubin levels more than twice the upper limit of normal).
* Psychological and cognitive disorders; dementia; major depression.
* Circadian rhythm disorders such as chronic fatigue syndrome and drowsiness.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-01-17 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 3 days postoperatively
  Postoperative pain will be assessed using the Visual Analogue Scale (VAS) at the following time points: upon arrival to the Post-Anesthesia Care Unit (PACU), and at 1, 2, 4, 6, 8, 12, and 24 hours, as well as at 12 and 24 hours on postoperative days 2 and 3.

SECONDARY OUTCOMES:
Incidence of postoperative anxiety | 3 days postoperatively
  Postoperative anxiety will be assessed using the Hospital Anxiety and Depression Scale (HADS) at the following time points:
  * 2, 6, and 24 hours on postoperative day 1,
  * 12 and 24 hours on both postoperative days 2 and 3.
  According to the HADS scoring system:
  1. A score of 0-7 is considered normal,
  2. 8-10 indicates a borderline case,
  3. 11-21 reflects abnormal anxiety. This assessment timeline enables comprehensive monitoring of anxiety levels during the critical early postoperative period
Postoperative analgesic consumption | 3 days postoperatively
  Postoperative analgesic consumption will be recorded.
Postoperative sleep quality | 3 days postoperatively
  Postoperative sleep quality will be recorded before surgery and every day for three days postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.